CLINICAL TRIAL: NCT03273218
Title: Effectiveness of the Tiger Catheter as a Simple Multipurpuse Catheter in Transradial Coronariography: Randomized Comparerd to Judkins Catheters
Brief Title: Effectiveness of the Tiger Catheter on Transradial Coronariography: Randomized Compared to JudKins cathETers
Acronym: TICKET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marcelo Alberto OLIVA (Other)
Responsible Party: Sponsor-Investigator, Marcelo Alberto OLIVA, interventional cardiologist, Hospital San Roque
Organization: Hospital San Roque (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HospitalSR
Record Dates: First submitted 2017-08-19; First posted 2017-09-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2017-08

CONDITIONS: Acute Coronary Syndrome
Keywords: coronary angiography; diagnosctic transradial catheter; transradial catheter
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Tiger catheter (Experimental): Tiger simple multipurpose catheter compared to Judkins catheters
  Interventions: Device: Tiger catheter
- Judkins catheter (Active Comparator): Judkins right and judkins left catheter
  Interventions: Device: Judkins catheter

INTERVENTIONS:
Device: Tiger catheter
  Other Names: Tiger
  Arms: Tiger catheter
Device: Judkins catheter
  Other Names: judkins right; judkins left
  Arms: Judkins catheter

SUMMARY:
The aim of this study was to assess effectiveness and safety of Tiger (5Fr) vs Judkins (5Fr) catheters, in coronariography via the right transradial approach.

This was a prospective, randomized, study of paralled design. Consecutive patients with acute coronary syndrome (ACS), eligible for coronary angiography, was randomized after successuful cannulation of right artery and informed consent to either Tiger or Judkins catheters.

DETAILED DESCRIPTION:
analyzed a total of 120 consective diagnostic coronary angioggraphy cases from the right radial approach. Of these 60 cases were performed with single catheter (Tiger) and 60 cases were performed with conventional catheters (Judkins). The patients of both group were overall well balanced for gender, age, risk factors, height, weight and body surface area. Diagnostic angiograms were successfully achieved in all cases via the radial approach.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* indication for coronary angiography

Exclusion Criteria:

* negative Allen´s test
* Chronic renal failure (to preserve the right radial artery for potencial arteriovenous shunting)
* Hemodynamic instability
* coronary artery bypass grafting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07-20 (Actual); Study Completion 2016-07-20 (Actual)

PRIMARY OUTCOMES:
Produce time for the coronary angiography | Day 0 (corresponding to time point of produce) assessed by intention - to - tresat analysis (IIT)
  Produce time (min) was defined as the time from the insertion of the first diagnostic coronary catheter in the sheath to the exist of the las diagnostic catheter the sheath.

SECONDARY OUTCOMES:
Fluoroscopy time | Day 0 (corresponding to time point of produce)
  Fluoroscopy time (min)was defined as fluoroscopy time during the procedure (between groups)
Contrast Volume used | Day 0 (corresponding to time point of produce)
  contrast volume used (ml) was defined as the contrast volume between groups used for completion of coronary angiogram
Radial artery Spasm | Day 0 (corresponding to time point of produce). The radial artery spasm was recorded like YES or NOT.(registry did by nurse from beginning to end of coronary angiography)
  Radial artery Spasm was defined as the discomfort or pain in the arm, between groups

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo OLIVA, MD, Principal Investigator — Hospital San Roque
Locations (1):
- Hospital San Roque, Córdoba, Argentina

IPD SHARING:
Plan to Share IPD: No
The aim of this study was to assess effectiveness and safety of Tiger vs Judkins catheters, in coronary angiography.

DOCUMENTS (1):
  • Study Protocol (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT03273218/Prot_000.pdf